CLINICAL TRIAL: NCT07211191
Title: Comparison of Functional Vestibulo-Ocular Reflex and Cognitive Functions in E-Athletes and Non-Athletes: A Cross-Sectional Case-Control Study
Brief Title: Comparison of Vestibulo-Ocular Reflex and Cognitive Functions in E-Athletes and Non-Athletes
Status: Completed | Type: Observational
Sponsor: Yusa Basoglu (Other)
Collaborators: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor-Investigator, Yusa Basoglu, Assistant Professor of Audiology, Medipol University
Organization: Medipol University (Other)
Other Study IDs: IMU-EC-855-2021; Istanbul Medipol University (Other: Istanbul Medipol University Ethics Committee Decision No: 855/2021)
Record Dates: First submitted 2025-09-22; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Vestibulo-Ocular Reflex; Esports Participation; Cognitive Functioning
Keywords: Esports; E-Athletes; Stroop Test; Corsi Block-Tapping Test; Functional Head Impulse Test (F-HIT); Dynamic Visual Acuity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- E-Athletes: Healthy volunteers aged 17-27 years with at least 4 years of competitive esports experience and a minimum of 20 hours per week of training. All had normal or corrected-to-normal vision, normal Montreal Cognitive Assessment (MoCA) scores, and no neurological or psychiatric disorders or neck movement limitations. Participants were adaptable to cognitive and vestibular testing.
- Non-Athlete Controls: Healthy volunteers aged 17-27 years with no prior competitive esports or organized sports training. All had normal or corrected-to-normal vision, normal Montreal Cognitive Assessment (MoCA) scores, and no neurological or psychiatric disorders or neck movement limitations. Participants were adaptable to cognitive and vestibular testing.

SUMMARY:
This study aims to compare cognitive functions and functional vestibulo-ocular reflex (VOR) between e-athletes and non-athletes. Participants aged 17-27 years will complete the Stroop Test, Corsi Block-Tapping Test, and Functional Head Impulse Test (F-HIT) during a single baseline session. Cognitive measures will include attention, response inhibition, and visuospatial memory, while F-HIT will assess dynamic gaze stability. The study uses a cross-sectional design to explore potential differences between groups. Findings are expected to provide preliminary evidence on whether competitive gaming is associated with cognitive advantages or vestibular adaptations.

DETAILED DESCRIPTION:
Esports requires rapid visuomotor coordination, attentional control, and working memory. While traditional sports have been extensively studied in relation to cognitive and vestibular performance, limited evidence exists regarding esports. Some studies suggest that video gaming may improve executive function, visuospatial memory, and processing speed, whereas others have reported impairments in response inhibition. In addition, the potential effects of esports on vestibulo-ocular reflex (VOR) function, which is essential for gaze stability during head movements, remain largely unexplored.

This cross-sectional study is designed to compare cognitive and vestibular performance between esports athletes and non-athlete controls. Participants include young adults with and without at least four years of competitive gaming experience. Cognitive abilities are assessed with the Stroop Test, which measures selective attention, inhibition, and processing speed, and the Corsi Block-Tapping Test, which evaluates visuospatial short-term and working memory. Vestibular performance is assessed with the Functional Head Impulse Test (F-HIT), which measures dynamic visual accuracy during passive head impulses in horizontal and vertical planes.

The primary outcome is Stroop Test Part V completion time under interference conditions. Secondary outcomes include Stroop errors and corrections, forward and backward Corsi spans, and F-HIT percent correct answers. By integrating cognitive and vestibular assessments, this study aims to provide preliminary evidence on whether intensive esports participation is associated with cognitive advantages, vestibular adaptations, or both. The findings may contribute to a better understanding of the health and performance characteristics of esports athletes and guide the development of evidence-based training strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age between 17 and 27 years
* Normal or corrected-to-normal vision
* Montreal Cognitive Assessment (MoCA) score within normal limits
* No neurological or psychiatric disorder
* No neck movement restriction
* Ability to adapt to cognitive and vestibular tests
* For e-athlete group: ≥4 years of esports experience and ≥20 hours per week of training
* For control group: No prior competitive esports or organized sports training

Exclusion Criteria:

* Hearing loss or tinnitus affecting functional performance
* History of dizziness within the last 3 months
* Active or diagnosed migraine with vestibular involvement
* Benign paroxysmal positional vertigo (BPPV)
* History of head trauma
* Systemic or neurological diseases affecting cognitive or vestibular function
* Visual impairments not corrected with glasses or lenses

Ages: 17 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy young adults (17-27 years), including 18 esports athletes and 18 age-matched non-athlete controls, recruited from a university esports center and surrounding community.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Stroop Test Part V Completion Time (seconds) | Day 1 (Baseline, during a single test session)
  Completion time on Stroop Part V and errors on Part IV/V, indexing selective attention and inhibition. Participants are shown color-word stimuli and must name ink colors as quickly and accurately as possible.

SECONDARY OUTCOMES:
Stroop Test Part IV Errors (number of incorrect responses) | Day 1 (Baseline, during a single test session).
  Number of errors on Stroop Part IV, reflecting selective attention and inhibitory control. Participants are asked to state the ink color of incongruent color-word stimuli. Fewer errors indicate better performance.
Stroop Test Part IV Corrections (number of corrected errors) | Day 1 (Baseline, during a single test session).
  Description: Number of self-corrections in Stroop Part IV, reflecting cognitive control. Participants can correct verbal mistakes during the task; higher correction counts indicate reduced automatic inhibition.
Corsi Block-Tapping Test - Forward Span (maximum sequence length) | Day 1 (Baseline, during a single test session).
  Short-term visuospatial memory capacity. Participants are shown sequences of blocks tapped by the examiner and must reproduce the same order. Higher span indicates better memory.
Corsi Block-Tapping Test - Backward Span (maximum sequence length) | Day 1 (Baseline, during a single test session).
  Visuospatial working memory capacity. Participants are shown sequences of blocks tapped by the examiner and must reproduce them in reverse order. Higher span indicates better working memory.
Functional Head Impulse Test (F-HIT) Percent Correct Answers (%CA) | Day 1 (Baseline, during a single test session).
  Accuracy in identifying optotypes presented during rapid passive head impulses in horizontal, RALP, and LARP planes (3,000-6,000°/s²). Higher %CA indicates better functional vestibulo-ocular reflex.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, BEYKOZ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
he datasets generated and analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Olcek G, Basoglu Y, Basoglu I, Tomac S. Comparison of functional vestibulo-ocular reflex and cognitive functions in e-athletes and non-athletes. BMC Sports Sci Med Rehabil. 2026 Jan 27. doi: 10.1186/s13102-026-01546-7. Online ahead of print. PMID 41593662